CLINICAL TRIAL: NCT00057239
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study Evaluating the Efficacy, Safety and Tolerability of Two Doses (20mg and 60mg) of a Once-Daily Oral Formulation of GW353162 in Subjects With Major Depressive Disorder for a Treatment Period of Eight Weeks
Brief Title: An 8 Week Depression Study In Adults Diagnosed With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHB20001
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: GW353162; Major Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — radafaxine

INTERVENTIONS:
Drug: Radafaxine

SUMMARY:
A Placebo Controlled Study Evaluating Efficacy, Safety and Tolerability of Radafaxine in Patients with Major Depressive Disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD)
* Duration of current depressive episode 12 weeks - 24 months
* Patients can read and write at a level sufficient to provide a signed consent
* If female, patients must be practicing an acceptable method of birth control

Exclusion Criteria:

* Patients have other psychiatric disorders that would affect patient's response to treatment
* Patients have not responded to two or more adequate courses of antidepressant therapy
* Patients cannot be currently abusing illicit drugs or alcohol
* Patients are not currently receiving psychotherapy
* Patients have received electroconvulsive therapy within 6 months prior to screening
* Patients are pregnant or lactating

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 546
Dates: Start 2003-03; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score after 8 weeks of treatment | 8 Weeks

SECONDARY OUTCOMES:
Change in the MADRS score at other timepoints; change in Clinical Global Impression; percentage of remitters and responders based on the MADRS; change in disability, motivation, energy and pain;incidence of adverse events over course of study. | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, M.D., Study Director — GlaxoSmithKline
Locations (28):
- United States (28):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Farmington, Connecticut
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Edwardsville, Illinois
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, Farmington Hills, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, Kenilworth, New Jersey
  - GSK Investigational Site, Lawrence, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Conshohocken, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Woodstock, Vermont
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Brown Deer, Wisconsin